CLINICAL TRIAL: NCT06001437
Title: CTN-0126 Following Outcomes Remotely Within Addiction Recovery Domains
Brief Title: Following Outcomes Remotely Within Addiction Recovery Domains
Acronym: FORWARD
Status: Recruiting | Type: Observational
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, McHugh, R. Kathryn, Associate Professor, Mclean Hospital
Other Study IDs: 2023P000766; 3UG1DA015831-21S4 (NIH)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to describe outcome of people with opioid use disorder over the long-term by collecting monthly and yearly data on their recovery. Adults with opioid use disorder who participate will complete surveys monthly online and once per year by phone about their substance use, mental health, treatment involvement and functioning. The goal of this study is to better understand how people with opioid use disorder recover over time to improve intervention for this group.

DETAILED DESCRIPTION:
This is a longitudinal follow-up study that will collect yearly outcomes data on adults with opioid use disorder (OUD) who participated one of two prior clinical trials in the NIDA Clinical Trials Network. This longitudinal, observational study will entail annual phone and online assessments of domains of interest (e.g., substance use, treatment engagement) as well as monthly assessments that are distributed via text messaging and email to be completed electronically by the participant. No participant randomization will occur for this study, and study data will be considered observational in nature. We aim to characterize the long-term course of OUD and to evaluate the long-term course and recovery of OUD.

ELIGIBILITY:
Inclusion Criteria:

1. Be an enrolled participant in one of two applicable clinical trials and be no longer than 24 months after the final expected assessment for that trial.
2. Be willing and able to provide locator information for survey distribution (mobile number and/or email address).
3. Be willing to allow the linkage of prior clinical trial study data to the current study record.

Exclusion Criteria:

1. Unable to understand or communicate to complete consent or study assessments.
2. Are currently in jail, prison or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities.
3. Other factors that would cause harm or increased risk to the participant or close contacts or preclude the participant's full adherence with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with opioid use disorder who have previously participated in one of two applicable opioid use disorder clinical trials in the NIDA Clinical Trials Network.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-09-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Opioid Use | 12 months
  Count of months of opioid use.
Engagement in Treatment | 12 months
  Count of months engaged in treatment for opioid use disorder

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No